CLINICAL TRIAL: NCT01757353
Title: Detroit Area Study of College Student Lifestyles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Tim Bogg, Ph.D., Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R00AA017877 (NIH)
Record Dates: First submitted 2012-12-18; First posted 2012-12-28 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Excessive Alcohol Consumption

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Self-directed: Information only (Active Comparator): Participants in this arm will complete a baseline assessment, followed by a 50-minute brief motivational interview (the Brief Alcohol Screening and Intervention for College Students; BASICS) 10-14 days after the initial assessment. Participants in this arm will complete follow-up assessments at approximately 3 and 9 months.
  Interventions: Behavioral: Self-directed: Information only
- BASICS motivational interview (Active Comparator): Participants in this arm will complete a baseline assessment, immediately after which they will be administered alcohol-related informational sheets. These participants will participate in follow-up assessment sessions at approximately 3 and 9 months.
  Interventions: Behavioral: BASICS motivational interview
- BASICS plus normative enhancement motivational interview (Experimental): Participants in this arm will complete a baseline assessment, followed by a 60-minute brief motivational interview (the Brief Alcohol Screening and Intervention for College Students, with a normative enhancement module) 10-14 days after the initial assessment. Participants in this arm will complete follow-up assessments at approximately 3 and 9 months.
  Interventions: Behavioral: BASICS plus normative enhancement motivational interview

INTERVENTIONS:
Behavioral: BASICS motivational interview
  Arms: BASICS motivational interview
Behavioral: BASICS plus normative enhancement motivational interview
  Arms: BASICS plus normative enhancement motivational interview
Behavioral: Self-directed: Information only
  Arms: Self-directed: Information only

SUMMARY:
The goal of this research study is to compare three harm reduction approaches for at-risk college student drinkers. One approach provides generic risk-related information after an initial interview/questionnaire assessment session. A second approach uses an established motivational interviewing framework (Brief Alcohol Screening and Intervention for College Students; BASICS) that provides personalized feedback in a follow-up session. A third approach also uses BASICS, but tests the utility of a personality-informed module for this approach that is informed by the social investment hypothesis.

DETAILED DESCRIPTION:
While individual difference factors, such as trait self-control and subjective college student role investment, appear to be important predictors of excessive alcohol consumption and related problems, these factors are not typically incorporated into indicated prevention strategies. Indicated prevention usually focuses on groups or individuals who already express some aspects of a health-related problem (e.g., heavy episodic drinking), or who, at the very least, exhibit markers of risk (e.g., early age of first drink) associated with the development of a health-related problem (Gordon, 1987). The primary aim of the current proposal is to incorporate a personality-informed module into an existing motivational interviewing framework for alcohol-related harm reduction and test its efficacy compared to an information-only approach (i.e., informational packet) and a conventional strategy for indicated prevention (i.e., Brief Alcohol Screening and Intervention for College Students, BASICS; Dimeff et al., 1999) that has provided evidence for reduced risk of alcohol-related problems in randomized controlled trials (Borsari & Carey, 2000; 2005).

Motivational interviewing is a common technique used to address ambivalence and/or resistance to behavioral change. Motivational interviewing is commonly used in the context of health-related behaviors, such as excessive alcohol consumption, where an individual might not have experienced any serious consequences (e.g., driving while intoxicated), but may still be at risk for problems (Miller & Rollnick, 2002). In motivational interviewing, a tone of collaboration and attentiveness is considered critical to the success of the interaction. The primary goal is to guide an individual toward increased motivation to change (and actual behavioral change) by being responsive to the desires and concerns of the individual as it relates to change, and by having an individual commit to even the most modest of change goals (e.g., consuming beverages with reduced alcohol by volume in situations that are known to be high-risk, rather than a favorite, higher alcohol-by-volume beverage). Motivational interviewing is well-suited to accommodate a personality-informed module for change due to its emphasis on an individual's unique profile of factors.

In BASICS, a harm reduction approach is used to inform the assessment and content of the initial assessment session, as well as the follow-up feedback session (Dimeff et al., 1999). Consistent with research showing there to be a continuum of problems for alcohol and other externalizing behaviors (Bogg & Finn, 2010; Krueger et al., 2002), the harm reduction approach emphasizes that any movement toward reduced risk and harm, regardless of its impact, is positive movement, even if a person might be farther along the continuum of harm (Marlatt, 1998). The current proposal seeks to test an augmentation of the harm reduction approach of BASICS with a normative enhancement approach derived from the social investment hypothesis of the Cumulative Continuity Model of personality development (Roberts & Caspi, 2003).

According to the social investment hypothesis, the process of commitment to normative roles, such as college student, is ''thought to exact a form of social control through the role demands embedded in these contexts that call on individuals to act with more responsibility and probity'' (Roberts & Caspi, 2003; p. 203). To the extent that further commitment, investment, and involvement in the college student role can be fostered, then a concomitant increase in trait self-control should be expected as well, independent of harm reduction effects. As suggested by the findings described above, the effect of increased subjective college student role investment could be to deflect a risky trajectory for alcohol-related problems - an effect that could be further amplified by corresponding increases in trait self-control. This normative enhancement (NE) approach is posited to be particularly useful for those individuals who do not recognize or are steadfastly resistant to even minor harm reduction efforts conveyed through the motivational interviewing framework of BASICS. The strategy of the normative enhancement approach is to capitalize on an individual's goals for involvement in roles - especially those roles, such as college student, which are nominally voluntary in nature.

ELIGIBILITY:
Inclusion Criteria:

* We initially screen anonymously on the telephone for the inclusion/exclusion criteria (see attached phone screen). The responses obtained from respondents are used only to determine if they meet study criteria. Their names and responses are not recorded and the information they provide is shredded when the screen is completed.

  * be currently enrolled in full-time university coursework
  * be between the ages of 18 and 23 years
  * understand and be able to respond to screening questions in English
  * be able to read at a Grade 6 level
  * have consumed at least 4 (for women) or 5 (for men) standard drinks at least two times in the past 30 days OR typically consume at least 3 (for women) or 4 (for men) standard drinks on a drinking occasion
  * meet at least one of the DSM-IV diagnostic criteria for alcohol dependence OR score 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT

Exclusion Criteria:

* not have major cognitive impairments (i.e., assessed by whether they can understand and respond adequately to all screening questions)
* not have any history of traumatic brain injury. Subjects also are excluded if they report a history of any serious head injury.
* not have a history of psychotic symptoms or Bipolar Disorder
* not be taking medications for cancer, AIDS treatment, or epilepsy
* not be taking other medications that will affect behavior, such as major tranquilizers or antipsychotics
* not currently receiving voluntary or mandated counseling or treatment for substance use

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Past 30-day typical weekly alcohol consumption, as well as peak alcohol drinking episodes. From this information, past 30-day typical and peak blood alcohol content can be calculated. | up to 9 months
  This measure is assessed using a structured interview.
Young adult alcohol consequences questionnaire | up to 9 months
  This instrument assesses the co-occurrence of behavioral problems and alcohol consumption, including physical, social, performance, and risk-related behaviors and outcomes.
Hypothetical role-based decisions-to-drink questionnaire | up to 9 months
  Four hypothetical college student drinking scenarios that vary in rewarding and punishing role-related information assess decisions to attend, to drink, and how much alcohol would be consumed.

SECONDARY OUTCOMES:
Subjective college student role investment questionnaire | Baseline, 3, 9 months
  This scale assesses involvement, responsibility, importance, and investment in education and the college student role.
Trait self-control questionnaire | Baseline, 3, 9 months
  This scale assesses general dispositional tendencies for planning, thinking before acting, and impulse control

OTHER OUTCOMES:
Readiness to change drinking patterns questionnaire | Baseline, 3, 9 months
  This questionnaire assesses an individual's stage of motivation to enact alcohol-related behavioral change.
Comprehensve effects of alcohol questionnaire | Baseline, 3, 9 months
  This questionnaire assesses positive and negative drinking expectancies.
Alcohol perceived risks questionnaire | Baseline, 3, 9 months
  This questionnaire assesses a college student's perception of various risks and outcomes associated with alcohol consumption.
Drinking norms rating form | Baseline, 3, 9 months
  This questionnaire assesses a college student's perceptions of what is typical for the alcohol consumption patterns of most college students.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bogg, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Bogg T, Finn PR. A self-regulatory model of behavioral disinhibition in late adolescence: integrating personality traits, externalizing psychopathology, and cognitive capacity. J Pers. 2010 Apr;78(2):441-70. doi: 10.1111/j.1467-6494.2010.00622.x. PMID 20433626
- [Background] Borsari B, Carey KB. Two brief alcohol interventions for mandated college students. Psychol Addict Behav. 2005 Sep;19(3):296-302. doi: 10.1037/0893-164X.19.3.296. PMID 16187809
- [Background] Borsari B, Carey KB. Effects of a brief motivational intervention with college student drinkers. J Consult Clin Psychol. 2000 Aug;68(4):728-33. PMID 10965648
- [Background] Dimeff, L. A., Baer, J. S., Kivlahan, D. R., & Marlatt, G. A. (1999). Brief alcohol screening and intervention for college students: A harm reduction approach. New York: Guilford Press.
- [Background] Gordon, R. (1987). An operational classification of disease prevention. In J. A. Steinberg & M. M. Silverman (Eds.), Preventing mental disorders: A research perspective (DHHS Publication No. [ADM] 87-1492, pp. 20-26). Rockville, MD: National Institute of Mental Health.
- [Background] Krueger RF, Hicks BM, Patrick CJ, Carlson SR, Iacono WG, McGue M. Etiologic connections among substance dependence, antisocial behavior, and personality: modeling the externalizing spectrum. J Abnorm Psychol. 2002 Aug;111(3):411-24. PMID 12150417
- [Background] Marlatt, G. A. (1998). Harm reduction: Pragmatic strategies for managing high-risk behaviors. New York: Guilford Press.
- [Background] Miller, W. R., & Rollnick, S. (2002). Motivational interviewing: Preparing people for change (2nd ed.). New York: Guilford Press.
- [Background] Roberts, B. W. & Caspi, A. (2003). The cumulative continuity model of personality development: Striking a balance between continuity and change in personality traits across the life course. In R.M. Staudinger & U. Lindenberger (Eds.), Understanding human development: Lifespan psychology in exchange with other disciplines (pp. 183-214). Dordrecht, NL: Kluwer Academic Publishers.